CLINICAL TRIAL: NCT04632381
Title: A Phase 1b, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Trial of Intravenous Zotatifin in Adults With Mild or Moderate Coronavirus Disease 2019 (COVID-19)
Brief Title: Intravenous Zotatifin in Adults With Mild or Moderate COVID-19
Acronym: PROPEL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Effector Therapeutics (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: eFT226-0003
Record Dates: First submitted 2020-11-12; First posted 2020-11-17 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Corona Virus Infection
Keywords: COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 3:1 to receive zotatifin or placebo in 3 cohorts of 12 patients each. Cohorts will be sequentially enrolled at progressively higher zotatifin dose levels: 0.01, 0.02, or 0.035 mg/kg.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Matching placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Active Arm, Zota Cohort 1 (Active Comparator): 0.01 mg/kg zotatifin
  Interventions: Drug: Zotatifin
- Active Arm, Zota Cohort 2 (Active Comparator): 0.02 mg/kg zotatifin
  Interventions: Drug: Zotatifin
- Active Arm, Zota Cohort 3 (Active Comparator): 0.035 mg/kg zotatifin
  Interventions: Drug: Zotatifin
- Placebo (Placebo Comparator): 5% dextrose injection, USP
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zotatifin — Zotatifin is a potent and sequence-selective inhibitor of eukaryotic translation initiation factor (eIF) 4A1-mediated translation that imparts its regulation through a reversible enhancement of eIF4A1 binding to RNAs (ribonucleic acids) with specific polypurine motifs within the 5'-untranslated region (UTR).
  Other Names: Zota
  Arms: Active Arm, Zota Cohort 1; Active Arm, Zota Cohort 2; Active Arm, Zota Cohort 3
Drug: Placebo — 5% dextrose injection, USP
  Other Names: PBO
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability, the antiviral activity, and plasma pharmacokinetics (PK) of zotatifin administered intravenously (IV) to adults with mild or moderate COVID-19.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, dose-escalating study will evaluate the safety and efficacy of zotatifin administered IV to adults with mild or moderate COVID 19.

Patients will be randomized to receive zotatifin or placebo in 3 cohorts of 12 patients each. Cohorts will be sequentially enrolled at progressively higher zotatifin dose levels. Study drug will not be administered to patients who are hospitalized. The second dose of study drug will not be administered should a patient progress from mild or moderate COVID-19 to severe COVID-19 prior to or on Day 8. Patients will assess and record their symptoms daily through Day 22 and at follow up (30 days after last infusion) (or at the early termination visit [if conducted]) in a paper patient diary using the WHO 9-point ordinal scale for clinical improvement. Other safety and efficacy measures will be assessed according to the Schedule of Procedures on Days 1, 4, 8, 10, 15 (end of treatment visit), and 22, and at follow up (30 days after last infusion). On non-dosing days, study visits will be conducted as home health visits, except for the follow-up visit, which will be conducted as a telephone visit.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided informed consent and any authorizations required by local law;
2. Is a male or female patient ≥18 and <65 years of age;
3. Has a laboratory-documented positive test for SARS CoV 2 infection as determined by local laboratory using a standard, Food and Drug Administration (FDA)-approved viral RNA or viral antigen assay from any oral or respiratory sample collected within 48 hours of randomization;
4. Has at least 2 symptoms associated with COVID-19 (fever or chills, cough, shortness of breath or difficulty breathing on exertion, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, or diarrhea) starting no more than 5 days prior to randomization and has mild or moderate disease at screening and at time of randomization, defined as the following:

   * Mild COVID-19

     * Positive testing by standard reverse transcriptase polymerase chain reaction (RT-PCR) assay or equivalent test;
     * Symptoms of mild illness with COVID-19 that could include fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, without shortness of breath or dyspnea; and
     * No clinical signs indicative of moderate, severe, or critical severity;
   * Moderate COVID-19

     * Positive testing by standard RT-PCR assay or equivalent testing;
     * Symptoms of moderate illness with COVID-19, which could include any symptom of mild illness or shortness of breath with exertion;
     * Clinical signs suggestive of moderate illness with COVID-19, such as respiratory rate ≥20 breaths per minute, saturation of oxygen (SpO2) >93% on room air at sea level, heart rate ≥90 beats per minute; and
     * No clinical signs indicative of severe or critical severity;
5. Has adequate hepatic function during screening, defined as the following:

   * Serum alanine aminotransferase ≤3 × upper limit of normal (ULN);
   * Serum aspartate aminotransferase ≤3 × ULN; and
   * Serum bilirubin (total) ≤1.5 × ULN (unless due to Gilbert's syndrome or hemolysis);
6. Has adequate bone marrow function during screening, defined as the following:

   * Absolute neutrophil count ≥1.0 × 10 9/L;
   * Platelet count ≥75 × 109/L; and
   * Hemoglobin ≥90 g/L (9.0 g/dL or 5.6 mmol/L);
7. Has adequate renal function during screening, defined as measured or estimated glomerular filtration rate ≥60 mL/min, calculated by the Cockcroft-Gault formula using actual body weight;
8. Female patients of childbearing potential must meet all of the following criteria:

   * Is not pregnant (confirmed via a negative urine pregnancy test);
   * Is not breastfeeding; and
   * Is willing to use a protocol-recommended method of contraception or willing to abstain from heterosexual intercourse from the start of blinded study drug until at least 90 days after the last dose of blinded study drug; Note: A female patient is considered to be of childbearing potential unless she has had a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy; has medically documented ovarian failure (with serum estradiol and follicle-stimulating hormone levels within the institutional laboratory postmenopausal range and a negative serum or urine β-human chorionic gonadotropin); or is menopausal (age ≥55 years with amenorrhea for ≥6 months).
9. Male patients who can father a child must meet all of the following criteria:

   * Is willing to use a protocol-recommended method of contraception or willing to abstain from heterosexual intercourse with females of childbearing potential from the start of blinded study drug until at least 90 days after the last dose of blinded study drug; and
   * Is willing to refrain from sperm donation from the start of blinded study drug until at least 90 days after the last dose of blinded study drug; Note: A male patient is considered able to father a child unless he has had a bilateral vasectomy with documented aspermia or a bilateral orchiectomy.
10. Is willing to comply with the scheduled visits, drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions; and Note: Psychological, social, familial, or geographical factors that may preclude adequate study participation should be considered.
11. In the judgment of the Investigator, participation in the protocol offers an acceptable benefit to risk ratio when considering current disease status, medical condition, and the potential benefits and risks of alternative treatments for the patient's disease.

Exclusion Criteria:

1. Is hospitalized for COVID-19;
2. Has dyspnea at rest or while talking, or has signs and symptoms of overt or impending respiratory failure;
3. Has significant cardiovascular disease, defined by myocardial infarction, arterial thromboembolism, or cerebrovascular thromboembolism, within 3 months prior to randomization; symptomatic dysrhythmias or unstable dysrhythmias requiring medical therapy; angina requiring therapy; symptomatic peripheral vascular disease; New York Heart Association Class 3 or 4 congestive heart failure; ≥Grade 3 hypertension (diastolic blood pressure ≥100 mmHg or systolic blood pressure ≥160 mmHg); or history of congenital prolonged QT syndrome;
4. Has a history of chronic obstructive pulmonary disease or bronchial asthma requiring continuous treatment and/or intermittent or continuous oxygen within the 90 days prior to screening; Note: Intermittent use of a β2-agonist inhaler is allowed.
5. Has evidence of an ongoing or systemic bacterial, fungal, or viral infection (including upper respiratory tract infections) other than SARS-CoV-2 infection, recurrent or repeat SARS CoV 2 infection, or history of incompletely treated tuberculosis (TB) and/or suspected or known extrapulmonary TB; Note: Patients with localized fungal infections of the skin or nails are eligible. Patients may be receiving topical antifungals. Systemic administration of azole antifungals is prohibited (see Section 5.6).
6. Has significant infiltrates (involving >50% of lung parenchyma) on an optional standard of care chest X-ray or other lung imaging exam within 1 week of screening;
7. Has known significant electrocardiogram abnormalities at screening, including unstable cardiac arrhythmia requiring medication, left bundle branch block, second-degree atrioventricular (AV) block type II, third-degree AV block, ≥Grade 2 bradycardia, or QTcF >450 msec for men or >470 msec for women;
8. Has type 1 diabetes mellitus or type 2 diabetes mellitus;
9. Has a body mass index (BMI) >30 kg/m2;
10. Has received a live vaccine within 30 days prior to randomization;
11. Has had major surgery within 4 weeks (inclusive) prior to randomization;
12. Has had prior solid organ or bone marrow progenitor cell transplantation;
13. Has a malignant tumor (excluding a malignant tumor cured with no recurrence in the past 2 years, completely resected basal cell and squamous cell carcinoma of the skin, and completely resected carcinoma in situ of any type);
14. Has had prior high-dose chemotherapy requiring stem cell rescue;
15. Has a history of or active uncontrolled systemic or local autoimmune disorders or other conditions that might impair or compromise the immune system;
16. Has ongoing immunosuppressive therapy, including systemic corticosteroids; Note: At screening and during study participation, patients may be using systemic corticosteroids (doses ≤10 mg of prednisone or equivalent) or topical or inhaled corticosteroids.
17. Has ongoing use of a therapeutic anticoagulant or history of bleeding disorder;
18. Has ongoing use or plans to use antivirals against COVID-19;
19. Has used a moderate or strong inhibitor or inducer of CYP3A4 within 7 days prior to randomization or is expected to require use of a moderate or strong CYP3A4 inhibitor or inducer during study participation;
20. Has previously received investigational product in a clinical study within 30 days or within 5 elimination half-lives (whichever is shorter) prior to randomization or is planning to take part in another therapeutic clinical study while participating in this study; Note: Participation in observational studies is allowed.
21. Has a known history of HIV or hepatitis B virus, or active hepatitis C virus infection;
22. Has a known serious allergic reaction or hypersensitivity to components of zotatifin or placebo;
23. Has a history of drug abuse or use of narcotics in the past 2 years that in the opinion of the Investigator will preclude study compliance; or
24. Has any illness, medical condition, organ system dysfunction, or social situation, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to provide informed consent, adversely affect the patient's ability to cooperate and participate in the study, or compromise the interpretation of study results.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by the incidence of Treatment Emergent Adverse Events and Serious Adverse Events | 52 days
  Incidence of Treatment Emergent Adverse Events and Serious Adverse Events
Safety as assessed by the incidence of adverse events of special interest: | 52 days
  Adverse Events of Special Interest to be assessed:
  * Incidence of hospitalizations
  * incidence of cytokine release syndrome
  * hemophagocytic lymphohistiocytosis
  * acute respiratory distress syndrome
  * need for oxygen supplementation
Tolerability as assessed by changes in vital signs from baseline (Day 1) | 22 days
  Changes as assessed by respiration rate
Tolerability as assessed by changes in vital signs from baseline (Day 1) | 22 days
  Changes as assessed by heart rate
Tolerability as assessed by changes in vital signs from baseline (Day 1) | 22 days
  Changes as assessed by oxygen saturation
Tolerability as assessed by changes in vital signs from baseline (Day 1) | 22 days
  Changes as assessed by temperature
Tolerability as assessed by changes in vital signs from baseline (Day 1) | 22 days
  Changes as assessed by blood pressure
Tolerability as assessed by changes in clinical symptoms from baseline (Day 1) | 22 days
  Changes as assessed by physical exam
Tolerability as assessed by changes in clinical laboratory tests from baseline (Day 1) | 22 days
  Changes as assessed by serum chemistry
Tolerability as assessed by changes in clinical laboratory tests from baseline (Day 1) | 22 days
  Changes as assessed by hematology
Tolerability as assessed by changes in clinical laboratory tests from baseline (Day 1) | 22 days
  Changes as assessed by coagulation
Tolerability as assessed by changes in clinical laboratory tests from baseline (Day 1) | 22 days
  Changes as assessed by urinalysis

SECONDARY OUTCOMES:
Time to viral load undetectability; | 22 days
  Defined as the time to the first of 2 consecutive negative SARS-CoV-2 measurements assessed from swab specimen
Proportion of patients with SARS-CoV-2 viral load below the level of detectability; | 22 days
  Assessed by swab specimen
Mean change in SARS-CoV-2 viral load; | 22 days
  Assessed by swab specimen
The time to clinical resolution; | 52 days
  Defined as resolution of symptoms on the WHO 9-point ordinal scale for clinical improvement.
Zotatifin plasma concentrations | 15 days
  Concentrations at end of infusion, end of dosing interval, and on defined timepoint periods.

OTHER OUTCOMES:
Time to viral load undetectability | 22 days
  Time to the first of 2 consecutive negative SARS-CoV-2 measurements assessed from daily samples
Proportion of patients below the limit of detection | 22 days
  Assessed from daily saliva and anterior nasal samples
Mean change in viral load in saliva and nasal samples | 22 days
  Assessed from daily saliva and anterior nasal samples
Mean change in viral load in plasma | 22 days
  Assessed from plasma collected
Assessment and quantification of infectious virus | 22 days
  Assessed by plaque-based or comparable assay
Virus resistance | 22 days
  According Virus Analysis Plan
Change in the WHO 9-point ordinal scale for clinical improvement | 38 days
  Assessed in change from baseline to post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Warner, MD, Study Director — EFFECTOR Therapeutics, Inc.
Locations (4):
- United States (4):
  - Pinnacle Research Group, Anniston, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - Tampa General Hospital, Tampa, Florida
  - National Institute of Allergy and Infectious Diseases, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No
Following completion of the study, the data may be considered for publication.

REFERENCES:
- See also: Link to the study website; Propel Covid-19 Clinical Trial — https://www.yourpropelstudy.com/